CLINICAL TRIAL: NCT05549180
Title: Phase IV, Randomized, Multicenter and Double Clinical Trial Blind Designed to Assess Safety and Convenience of the Change From DTG/3TC to BIC/FTC/TAF in People With HIV, Good Virological Control and Neuropsychiatric Vulnerabilities: MIND Study
Brief Title: Phase IV, a Clinical Trial to Assess Safety and Convenience of the Change From DTG/3TC to BIC/FTC/TAF in People With HIV, Good Virological Control and Neuropsychiatric Vulnerabilities
Acronym: MIND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GESIDA 11920
Record Dates: First submitted 2022-06-01; First posted 2022-09-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: The drugs used will be drugs for commercial use that contain the active ingredients uses in this study:
  * Experimental regimen:
    * Bictegravir 50mg/ Emtricitabine 200mg/ Tenofovir alafenamide 25mg (combined in a single tablet marketed under the name of Biktarvy®). This regimen is given as 1 tablet once a day.
    * Placebo dolutegravir 50mg/ lamivudine 300mg (combined in a single tablet marketed under the name Dovato®). This regimen istake as 1 tablet once a day.
  * Control regimen:
    * Dolutegravir 50mg/ lamivudine 300mg (combined in a single tablet marketed under the name Dovato®). This regimen is administered as 1 tablet once a day.
    * Placebo bictegravir 50mg/ emtricitabine 200mg/ tenofovir alafenamide 25mg (combined in a single tablet marketed under the name of Biktarvy®). This regimen is given as 1 tablet once a day.
Who Masked: Participant, Investigator
Masking Description: The clinical trial is double blind.
  The only people who will know the arm that patient has been randomized, the participant will be responsible for the pharmacy in charge of dispensing treatment and a "non-blind" person designated by the promoter. The masking of study will only be open upon completion of the study or in the event that a participant developes a serious adverse event that requires knowing the treatment the patient is receiving participant for clinical management.
  If it is necessary a open blind premature manually, the investigator should contact the "non-blind" person designated by the the promoter by calling a phone number and indicating that they wish to break prematurely blinded a patient in the MIND study. After confirming that it is required to opening of the blind (because the condition described above occurs), the person "not blind" designated by the sponsor will indicate to the investigator the treatment arm that was receiving the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients received DTG/3TC + BIC/FTC/TAF placebo (Active Comparator): DTG 50 mg/3TC 300 mg 1 tablet per day + BIC 50 mg/ FTC 200 mg/ TAF 25 mg placebo 1 tablet per day
  Interventions: Drug: Dovato 50Mg-300Mg Tablet + Biktarvy placebo
- Patients received BIC/FTC/TAF + DTG/3TC placebo (Experimental): BIC 50 mg/ FTC 200 mg/ TAF 25 mg per day + DTG 50 mg/3TC 300 mg placebo1 tablet per day
  Interventions: Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet and Dovato placebo

INTERVENTIONS:
Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet and Dovato placebo — The patients randomized to experimental arm will be randomized to Biktarvy + Dovato placebo
  Arms: Patients received BIC/FTC/TAF + DTG/3TC placebo
Drug: Dovato 50Mg-300Mg Tablet + Biktarvy placebo — The patients randomized to comparador arm will be randomized to Dovato + Biktarvy placebo
  Arms: Patients received DTG/3TC + BIC/FTC/TAF placebo

SUMMARY:
In people infected with HIV, with suppressed HIV viral load and receiving treatment with DTG/3TC:

The change to BIC/FTC/TAF will decrease the development of adverse events of neuropsychiatric etiology.

The change to BIC/FTC/TAF may improve the patient´s tolerability and degree of acceptance and use of TAR.

DETAILED DESCRIPTION:
The clinical trial is designed to compare people with HIV and neuropsychiatric vulnerabilities, the safety and tolerability of switch to BIC/FTC/TAF versus continue on DTG/3TC.

The study includes the inclusion of 80 participants with HIV and who present among their personal history any of those established among the selection criteria (insomnia, anxiety or depression), agree to participate in the same The participants, after signing the informed consent and verifying the meeting of the selection criteria, they will be randomized to continue for 48 weeks with DTG/3TC + BIC/FTC/TAF placebo (arm 1) or switch to BIC/FTC/TAF + placebo DTG/3TC (arm 2).

All participants, except those who discontinue the study early, must to complete the same schedule of visits. It will be cause of early discontinuation loss to follow-up, withdrawal of consent, or development of any condition that requires discontinuation or change of assigned treatment.

During follow-up, the management of the basic neuropsychiatric pathology of each participant will be performed in accordance with normal clinical practice. In no case, the beginning, the change or the cessation of any pharmacological treatment or neuropsychiatric intervention should be affected by their participation in the study. If the situation arises where any participant developed a severe neuropsychiatric adverse effect (grade 3-4), two specialists in psychiatry experts in the management of patients with HIV would be responsible for evaluating them through the review of their medical history and an interview with the participant in person or via telematics. This evaluation will aim to confirm the relevance of the continuity of the patient in the study and the need for further preferential evaluation by psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years diagnosed with HIV by standard microbiological techniques
* Active antiretroviral treatment with DTG/3TC
* Last HIV viral load performed on the participant in the 6 months prior to the visit screening < 50 copies/mL. If the participant does not have an HIV viral load <50 cop/mL performed in the 14 days prior to the screening visit, it will be necessary to confirm at screening visit that the participant's HIV viral load is <50 cop/mL
* Prior clinical diagnosis, carried out by a qualified specialist physician, of any of the following pathologies: Insomnia Anxiety disorders Depressive disorders

Exclusion Criteria:

* Allergy or intolerance to any of the components of BIC/FTC/TAF
* History of active CNS infections
* Active psychosis or suicidal ideation
* Pregnant or lactating women, as well as women of childbearing age who do not commit to use at least two contraceptive methods
* Any clinical or laboratory condition that in the opinion of the investigator will prevent the participant to complete the study procedures
* Participant included in the neuroimaging substudy: Claustrophobia or presence of magnetizable body devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
The safety of switching to BIC/FTC/TAF versus continuing treatment with DTG/3TC. | 24-48 weeks
  Primary endpoint: Proportion of neuropsychiatric adverse effects grade 2-4 (defined using the AIDS Clinical Trials Group Adverse Events Grading Score11)
  Secondary endpoints:
  1. Proportion of grade 2-4 adverse effects (defined using the AIDS Clinical Trials Group Adverse Events Grading Score11)
  2. Proportion of ART discontinuations due to neuropsychiatric adverse effects.
  3. Proportion of ART discontinuations for any reason.

SECONDARY OUTCOMES:
The desirability of switching to BIC/FTC/TAF versus continuing treatment with DTG/3TC. | 24-48 weeks
  Primary endpoint: Changes in sleep quality estimated using the Pittsburgh Sleep Quality Questionnaire (PSQI)
  Secondary endpoints:
  1. Changes in mood estimated using the hospital scale of anxiety and depression (HADS)
  2. Changes in the scale of satisfaction with ART (ESTAR)
  3. Changes in the Spanish version of the MOS HIV quality of life questionnaire.
The efficacy of switching to BIC/FTC/TAF versus continuing treatment with DTG/3TC. | 24-48 weeks
  Primary endpoint: Percentage of participants with HIV viral load >50 copies/mL, according to the Snapshot algorithm of the "US Food and Drug Administration" (margin to demonstrate non-inferiority: 4%)
  Secondary edpoints:
  * 1)Proportion of participants with HIV viral load <50 copies/mL
    2) Proportion of participants with undetectable viral load.
    3) Proportion of patients with failure confirmed virology
    4) Percentage of patients with virological failure
    5) Proportion of participants experiencing blips during the study

OTHER OUTCOMES:
Exploratory outcome: Brain integrity and functionality before and after switching to BIC/FTC/TAF. | 48 weeks
  Primary endpoint: Changes in brain volumes
  Secondary endpoints:
  1. Changes in the levels of N-acetyl-aspartate, choline and myo-inositol at the frontal grey matter, frontal white matter, and basal ganglia
  2. Changes in the integrity of the white matter
  3. Changes in cerebral perfusion
  4. Changes in brain resting state

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - H. Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - CHUAC, A Coruña
  - Hospital de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Fundacion Hospital Alcorcón, Madrid
  - H. Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - H. Costa del Sol, Marbella
  - Hospital Son Llatzer, Palma de Mallorca
  - H. Univ. Virgen Macarena, Seville
  - H. Clinico Univ. Lozano Blesa, Zaragoza